CLINICAL TRIAL: NCT05345808
Title: Efficacy of Formulated Posterior Sub Tenon Triamcinolone in Macular Edema Secondary to Non-Ischemic Retinal Vein Occlusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Akram Fekry Elgazzar, Clinical Professor, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSTA in macular edema
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formulated Posterior Sub Tenon Triamcinolone (Other): All the eyes received single dose 40 mg of Triamcinolone Acetonide (TA) and VISCOAT which is 20 mg sodium chondroitin sulphate and 15 mg sodium hyaluronate (0.5 ml) through posterior subtenon route using NAGATA subtenon canula.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Triamcinolone Acetonide formulated with chondroitin sulfate and sodium hyaluronate

SUMMARY:
Retinal vein occlusion (RVO) is considered the second vascular disorder of the retina after diabetic retinopathy. Patients with RVO are at risk of the development of macular edema. Different treatment modalities for macular edema include LASER therapy, antivascular endothelial growth factor (VEGF), and triamcinolone.

Aim To detect the efficacy of formulated Triamcinolone Acetonide(TA) injection in the posterior subtenon space to manage macular edema secondary to non-ischemic RVOs, either central or branch.

ELIGIBILITY:
Inclusion Criteria:

* Diminution of vision due to macular edema secondary to non-ischemic retinal vein occlusions, either central or branch
* CMT ≥ 250 µ,
* Willing to participate in the study.

Exclusion Criteria:

* Unwilling to participate in the study
* Ischemic RVO
* previous laser treatment
* Glaucoma, macular ischemia, cataract, vitreous hemorrhage, and neovascularization of the iris
* patients with previous anti VEGFs or steroid injections or any eye surgery three months before the inclusion
* Cardiac co-morbidities result in significant hemodynamic changes
* Respiratory diseases need treatment with antibiotics
* Suffering from other chronic diseases as diabetes
* Patient with allergy from triamcinolone acetonide.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | at the base line
  Measured by snellen chart
Best corrected visual acuity | at 1st month
  Measured by snellen chart
Best corrected visual acuity | at 3rd month
  Measured by snellen chart
Best corrected visual acuity | at 6th month
  Measured by snellen chart
Central macular thickness | at 1st month
  Measured by Optical coherence tomography (OCT)
Central macular thickness | at 3rd month
  Measured by Optical coherence tomography (OCT)
Central macular thickness | at 6th month
  Measured by Optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Akram Fekry Elgazzar, Damietta, Egypt